CLINICAL TRIAL: NCT06488638
Title: Pilot Study of Nitrate-rich Beetroot Juice Supplementation in Patients With Idiopathic Pulmonary Fibrosis (IPF)
Acronym: BEET-IPF
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Southampton NHS Foundation Trust (Other)
Collaborators: NIHR Southampton Respiratory Biomedical Research Centre (Unknown); Asthma, Allergy and Inflammation Research (AAIR) Charity (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: RHMRESP0009
Record Dates: First submitted 2024-06-26; First posted 2024-07-05 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2024-07

CONDITIONS: Idiopathic Pulmonary Fibrosis; Interstitial Lung Disease
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis; Lung Diseases, Interstitial | interventions — Nitrates

STUDY DESIGN:
Intervention Model Description: placebo-controlled, double blind, randomised controlled trial
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Treatment period 1) nitrate-rich beetroot juice (70ml with approx. 400 mg nitrate) twice a day for 3 days
  Treatment period 2) placebo nitrate-depleted beetroot juice (70ml) twice a day for 3 days
  Interventions: Dietary Supplement: nitrate-rich beetroot juice (70ml with approx. 400 mg nitrate) twice a day for 3 days
- Group B (Placebo Comparator): Treatment period 1) placebo nitrate-depleted beetroot juice (70ml) twice a day for 3 days
  Treatment period 2) nitrate-rich beetroot juice (70ml with approx. 400 mg nitrate) twice a day for 3 days
  Interventions: Dietary Supplement: nitrate-rich beetroot juice (70ml with approx. 400 mg nitrate) twice a day for 3 days

INTERVENTIONS:
Dietary Supplement: nitrate-rich beetroot juice (70ml with approx. 400 mg nitrate) twice a day for 3 days — commercially available beetroot juice dietary nitrate supplement

SUMMARY:
Idiopathic pulmonary fibrosis (IPF) is a type of scarring (fibrotic) lung disease. Reduced exercise capacity is a key symptom experienced by patients. In previous research the investigators identified that an interval-based exercise programme led to significant improvements in exercise capacity (Wallis et al Antioxidants. 2023).

An unexpected finding was that in patients with IPF, exercise led to a reduction in blood nitrite concentrations an observation the investigators did not see in non-affected individuals. Research has identified that nitrite concentrations are expected to increase after exercise and the size of this increase is related to an individual's exercise capacity. There is also evidence from healthy individuals and patients with chronic obstructive pulmonary disease (COPD) that nitrate supplementation (a source of nitrite) improves response to exercise training. However, in both these groups an exercise-induced fall in blood nitrite concentrations has not been observed. Hence our finding of an exercise-induced fall in blood nitrite levels in IPF patients suggest that they may be especially sensitive to supplementation with nitrate, commercially available as nitrate-rich beetroot juice (NRBJ).

This current study investigates this in a pilot placebo-controlled, double-blind, randomised, cross-over study of NRBJ on exercise capacity in IPF patients.

Aims In patients with IPF

* Quantify the effect of nitrate supplementation on exercise capacity
* Determine the effect of nitrate supplementation on blood markers of nitric oxide production/metabolism.
* Determine the effect of nitrate supplementation on forearm blood flow. Sample size: n=8 IPF patients, aged 18-85years and medical research breathlessness scale 1-3 Intervention: 3-days (two-times daily) NRBJ or nitrate-depleted placebo juice (both commercially available) with subsequent constant-load exercise test (Primary outcome). Following at least 1 week wash-out period participants will cross-over and repeat.

A cohort (n=8) of age, sex-matched controls without IPF will be enrolled for comparison of forearm blood flow and pre-exercise venous blood samples for biomarkers comparison only.

Number of sites: 1

DETAILED DESCRIPTION:
Idiopathic pulmonary fibrosis (IPF) is the prototypic chronic progressive fibrotic interstitial lung disease (ILD). Progressive disease is characterised by breathlessness and exercise limitation and there is an unmet need for interventions which improve patient's quality of life. Increasing exercise intolerance in patients with ILD is associated with worsening quality of life and loss of independence. Pulmonary rehabilitation is recommended by the National Institute for health and Care Excellence (NICE) for patients with ILD, however individual responses to exercise training are variable and optimal training strategies are yet to be established.

In previous published research (Wallis et al. 2023. Antioxidants) the investigators studied the effect of an individually prescribed, interval-based aerobic exercise programme on redox status and functional capacity in patients with IPF. At baseline, IPF patients had evidence of increased oxidative stress. The individually prescribed exercise programme led to a significant increase in antioxidant buffering capacity together with clinically meaningful improvements in exercise capacity and medical research council (MRC) breathlessness score. Notably, the investigators also identified that in patients with IPF, exercise induced a significant fall in circulating nitrite concentrations, an effect potentiated by exercise training. In contrast, control individuals exhibited a post-exercise increase in nitrite concentrations due to shear stress-induced nitric oxide (NO)-synthase stimulation.

Nitric oxide (NO) physiology is strongly implicated in the physiology of exercise performance. In healthy individuals the delta of the post-exercise increase in circulating nitrite concentration positively correlates with peak exercise capacity and it has been identified that supplementation with nitrate significantly lowers the oxygen cost (oxygen uptake [V̇O2] required to perform a given work-rate) of submaximal exercise. Recent evidence from patients with COPD has identified that sustained supplementation with nitrate-rich beetroot juice augmented the effect of pulmonary rehabilitation compared to placebo (+30m in incremental shuttle walk test). However, in contrast to our findings in IPF, within these groups no underlying dysregulation in nitrite utilisation during exercise has been identified i.e. exercise induced nitrite decrease is not present. This suggests that patients with IPF may be exquisitely sensitive to benefit from nitrate (known to serve as a source of nitrite) during exercise, a non-pharmacologic intervention with potential rapid translation into clinical practice.

Hypothesis

Nitrate supplementation (in the form of nitrate-rich beetroot juice drink) significantly improves submaximal exercise capacity in patients with IPF.

Here the investigators test this hypothesis in this study by way of a pilot randomised controlled double-blind cross-over study of nitrate supplementation on submaximal exercise capacity in patients with IPF. Together with a nested mechanistic study investigating the effect of nitrate supplementation on systemic blood markers of nitric oxide production and metabolism as well as forearm blood flow.

Aims and Objectives

In patients with IPF

1. Quantify the effect of nitrate supplementation on submaximal exercise capacity (constant work-rate test).
2. Determine the effect of nitrate supplementation on markers of nitric oxide (NO) production and metabolism pre- and post-exercise.
3. Determine the effect of nitrate supplementation on forearm blood flow.
4. Assess the effect of nitrate supplementation of participants' perceptions of exercise and quality of life

Study Design and setting Up to 8 patients with IPF will be recruited to this single centre cohort cross-over double-blind designed pilot study at a large NHS Foundation trust teaching hospital. Ongoing interim analysis will be conducted throughout the study.

Intervention Participants will be randomly assigned to either 3-days (two times daily) of nitrate-rich beetroot juice drink (daily dose of nitrate 800mg nitrate) or nitrate-depleted juice placebo control drink of identical taste and colour (Treatment Period 1) immediately prior to constant-load exercise test (see intervention). Following a wash-out period of at least 1-week they will cross-over and repeat (Treatment Period 2).

Control Cohort:

A cohort (n=8) of age and sex-matched controls without IPF will be enrolled for comparison of forearm blood flow by venous occlusion plethysmography (VOP) and pre-exercise venous blood samples for biomarkers of NO metabolism and oxidative stress.

End points: Endurance time, adverse events. Number of sites: 1

ELIGIBILITY:
Cases Inclusion Criteria

1. Patients aged 18-85 years with a prior specialist multidisciplinary team diagnosis of idiopathic pulmonary fibrosis (IPF) based on current established consensus guidelines.
2. Medical Research Council (MRC) breathlessness grade 1-3
3. Judged clinically stable for 3 months prior to recruitment by the investigator.

Exclusion Criteria

1. Baseline spirometry with FEV1/FVC ratio < 0.7.
2. Neoplastic disease undergoing treatment or active follow up.
3. Presence of infection or exacerbation requiring hospitalization, within last 3 months.
4. Current tobacco smoker or use of nicotine containing vapes (within 3months)
5. Current use of ambulatory or long-term oxygen therapy (LTOT).
6. Peripheral oxygen saturations <85% during 6-minute walk-test.
7. Any condition which would prevent completion of cycle-ergometer testing, pulmonary function testing (PFT) or 6-minute walk testing as judged by the investigator.
8. Participation in a pulmonary rehabilitation (PR) program in the last 3 months.
9. Any condition excluding CPET based on the absolute contraindication as the ACCP/ATS guidelines 2003
10. Positive pregnancy test in females of childbearing age.
11. Symptomatic peripheral vascular disease

Controls Control Inclusion Criteria

1) Age and sex-matched to participants in the IPF cohort Control Exclusion Criteria

1. Inability to give informed written consent
2. Malignancy (except localized squamous or basal cell skin carcinoma) undergoing active investigation, treatment, or follow-up
3. Significant cardiorespiratory disease as judged by the investigator
4. Diabetes mellitus requiring treatment with pharmacology therapy
5. Current tobacco smoker or use of nicotine containing vapes (within 3months)
6. Symptomatic peripheral vascular disease

Ages: 28 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
endurance time | From end of treatment period 1 to end of treatment period 2 (minimum 10 days)
  fixed-load static cycle ergometry test

SECONDARY OUTCOMES:
plasma nitrate and nitrite concentrations | From end of treatment period 1 to end of treatment period 2 (minimum 10 days)
  venous blood samples
forearm blood flow | From end of treatment period 1 to end of treatment period 2 (minimum 10 days)
  venous occlusion plethysmography

CONTACTS AND LOCATIONS:
Overall Officials: Tim JM Wallis, MD, PhD, Study Chair — University Hospital Southampoton

IPD SHARING:
Plan to Share IPD: No